CLINICAL TRIAL: NCT00718692
Title: A Multi-centre, Single Intravenous Dose, Exploratory Dose-finding, Open Label Trial on the Safety and Efficacy of Sym001 in the Treatment of Immune Thrombocytopenic Purpura (ITP) in RhD Positive, Non-splenectomized Adult Subjects.
Brief Title: Open Label Trial on the Safety and Efficacy of Sym001 in the Treatment of Immune Thrombocytopenic Purpura (ITP)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Symphogen A/S (Industry)
Collaborators: Swedish Orphan Biovitrum (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Sym001-03; 2007-006081-15 (EudraCT Number)
Record Dates: First submitted 2008-07-18; First posted 2008-07-21 (Estimated); Last update posted 2019-01-30 (Actual); Status verified 2019-01

CONDITIONS: Immune Thrombocytopenic Purpura
Keywords: Idiopathic; ITP
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — rozrolimupab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Patients treated with Sym001
  Interventions: Drug: Sym001

INTERVENTIONS:
Drug: Sym001 — Each cohort will receive one single dose of Sym001 according the assigned dose level.

SUMMARY:
This trial is designed as a multi-centre, single-dose, exploratory dose-finding, open label trial evaluating the safety and efficacy of Sym001 in 4-9 consecutive cohorts. Subjects will receive a single IV dose of Sym001.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed presence of thrombocytopenia with platelet count < 30,000/mm3 at the pre-dose visit.
* History of isolated ITP
* RhD-positive serology.
* Previous treatment and response to first line therapy for ITP

Exclusion Criteria:

* Known clinical picture suggestive of other causes of thrombocytopenia, especially systematic lupus erythematosus,antiphospholipid syndrome, Evans syndrome, immunodeficiency states, lymphoproliferative disorders, liver disease,ingestion of drugs such as quinidine/quinine, heparin and sulfonamides and hereditary thrombocytopenia confirmed by relevant laboratory findings.
* Suspected infection with HIV, Hepatitis C, H. pylori.
* Clinical splenomegaly
* History of abnormal bone marrow examination.
* Ongoing haemorrhage corresponding to a grade 3 or 4 on the WHO bleeding scale.
* Underlying haemolytic condition
* History of splenectomy.
* Subject is pregnant, breast feeding or intends to become pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2008-07 (Actual); Primary Completion 2011-08 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of Adverse Events (AEs), including Serious Adverse Events (SAEs) | 6 weeks post dosing

SECONDARY OUTCOMES:
Measurements of platelet counts | From day 1 through week 6

CONTACTS AND LOCATIONS:
Overall Officials: Mario Von Depka Prondzinski, PD Dr., Principal Investigator — Werlhoff Institut Hannover, Germany; Ann Janssens, Dr., Principal Investigator — ZU Gasthuisberg, Leuven, Belgium; Javier Loscertales Pueyo, Dra, Principal Investigator — Hospital La Princesa, Madrid, Spain; Wieslaw Wiktor Jedrzrjczak, Prof., Principal Investigator — Katedra i klinika Hematologii, Warszawa, Poland; Andrei Cucucianu, Dr., Principal Investigator — Prof. Dr. Ion Chiricuta Oncology Institute, Cluj-Napoca, Romania; Marie Scully, Prof. Dr. MD, Principal Investigator — University College London Hospitals
Locations (59):
- United States (3):
  - Univ Nebraska Med Ctr. UNMC, 1005, Omaha, Nebraska
  - Hospital of the University of Pennsylvania, Site 1002, Philadelphia, Pennsylvania
  - 2085 Henry Tecklenburg Drive, 1001, Charleston, South Carolina
- Belgium (3):
  - Research Site 3203, Bruges
  - Research Site 3202, Leuven
  - Research Site 3201, Yvoir
- Germany (7):
  - Research Site 4906, 4907, Berlin
  - Research Site 4902, Cologne
  - Research Site 4903, Duisburg
  - Research Site 4905, Essen
  - Reseach Site 4908, Halle
  - Research Site 4901, Hanover
  - Research Site 4904, Regensburg
- India (7):
  - St. John's Medical College Hospital, 9106, Bangalore
  - MS Ramaiah Memorial Hospital, 9108, Bangalore
  - Narayana Hrudayalaya Hospitals, 9105, Bangalore
  - Columbia Asia Referral Hospital-Yeshwanthpur, 9101, Bangalore
  - Aysha Hospital Pvt. Ltd., 9109, Chennai
  - Apollo Hospital, 9104, Hyderabad
  - Kasturba Medical College Hospital, 9103, Udupi
- Israel (6):
  - Bnai-Zion Medical Center, 9721, Haifa
  - Rambam Medical Center, 9723, Haifa
  - The Edith Wolfson Medical Center, 9725, Holon
  - Western Galilee - Nahariya Hospital, 9722, Nahariya
  - Rabin Medical Center, 9724, Petah Tikva
  - Tel-Aviv Sourasky Medical Center, 9726, Tel Aviv
- Poland (7):
  - Research site 4801, Gdansk
  - Research Site 4806, Krakow
  - Research Site 4805, Lodz
  - Instytut Hematologii i Transfuzjologii, 4807, Warsaw
  - Research Site 4802, 4808, Warsaw
  - Research Site 4803, Warszava
  - Research Site 4804, Wroclaw
- Romania (4):
  - Brasov Country Hospital, 4002, Brasov
  - Institutul Clinic Fundeni, 4003, Bucharest
  - "Prof. Dr. Ion Chiricuta" Oncolgy Institute, 4001, Cluj-Napoca
  - Spitalul Clinic de Urgente Sfantu Spiridon, 4004, Iași
- Russia (4):
  - Regional Clinical Hospital of Nizhny Novgorod, 7003, Nizhny Novgorod
  - Saint Petersburg State Institution Of Healthcare, 7001, Saint Petersburg
  - Regional Clinical Hospital na MI Kalinin, 7005, Samara
  - State Healthcare Institution Tula Regional Clin. Hosp., 7002, Tula
- Serbia (3):
  - Clinical Center Nis 3802, Niš
  - Clinical center Vojvodina 3801, Novi Sad
  - Clinical Center Zemun 3803, Zemun
- Spain (5):
  - Reseach Site 3403, Barcelona
  - Hospital Gregorio Maranon, 3405, Madrid
  - Hospital La Princesa, 3404, Madrid
  - Research Site 3401, Madrid
  - Research Site 3402, Valencia
- Ukraine (5):
  - Cherkassy regional oncology center, 3906, Cherkassy
  - Gusak Academy of AMS Ukraine, 3905, Donetsk
  - Khmelnytskyi Regional Hospital, 3903, Khmelnytskyi
  - City Hospital #9 Kyiv Clinical Hospital, 3904, Kiev
  - Vinnytsya Regional Clinical Hospital, 3902, Vinnytsia
- United Kingdom (5):
  - St. James's University Hospital, 4403, Leeds
  - Hammersmith Hosptial, 4402, London
  - University College, 4401, London
  - Royal Victoria Infirmery, 4404, Newcastle upon Tyne
  - Singleton Hospital, 4405, Swansea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Robak T, Windyga J, Trelinski J, von Depka Prondzinski M, Giagounidis A, Doyen C, Janssens A, Alvarez-Roman MT, Jarque I, Loscertales J, Rus GP, Hellmann A, Jedrzejczak WW, Kuliczkowski K, Golubovic LM, Celeketic D, Cucuianu A, Gheorghita E, Lazaroiu M, Shpilberg O, Attias D, Karyagina E, Svetlana K, Vilchevska K, Cooper N, Talks K, Prabhu M, Sripada P, Bharadwaj TP, Naested H, Skartved NJ, Frandsen TP, Flensburg MF, Andersen PS, Petersen J. Rozrolimupab, a mixture of 25 recombinant human monoclonal RhD antibodies, in the treatment of primary immune thrombocytopenia. Blood. 2012 Nov 1;120(18):3670-6. doi: 10.1182/blood-2012-06-438804. Epub 2012 Aug 20. PMID 22915649